CLINICAL TRIAL: NCT03342040
Title: Randomized Clinical Trial: Transverse Abdominis Plane Block Versus no Block in Laparoscopic Ventral Hernia Repair
Brief Title: Transverse Abdominis Plane Block in Laparoscopic Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GEM Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GemHRC
Record Dates: First submitted 2017-09-29; First posted 2017-11-14 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Ventral Hernia
Keywords: TAP block; laparoscopic IPOM; post operative pain
MeSH Terms: conditions — Hernia, Ventral; Pain, Postoperative | interventions — Bupivacaine; Ropivacaine; Injections, Subcutaneous

STUDY DESIGN:
Intervention Model Description: Prospective double blinded balanced allocation, randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and assessors are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Experimental): Patients undergoing laparoscopic ventral hernia repair with TAP block with 0.2% ropivacaine under ultrasound guidance
  Interventions: Procedure: Laparoscopic ventral hernia repair with TAP block
- No TAP block (Active Comparator): Patients undergoing laparoscopic ventral hernia repair without TAP block
  Interventions: Procedure: Laparoscopic ventral hernia repair without TAP block

INTERVENTIONS:
Procedure: Laparoscopic ventral hernia repair with TAP block — Transverse abdominis plane block is given under ultrasound guidance during laparoscopic ventral hernia surgery
  Other Names: Bupivacaine 0.25% and Ropivacaine 0.2% subcutaneous injection
  Arms: TAP block
Procedure: Laparoscopic ventral hernia repair without TAP block — No block administered during Laparoscopic ventral hernia surgery
  Arms: No TAP block

SUMMARY:
The current study aims to determine if transverse abdominis plane block using local anesthetic agents (bupivacaine 0.25% + Ropivacaine 0.20%) decreases the post operative pain and helps in early mobilization or discharge from hospital in patients undergoing laparoscopic ventral hernia repair.

DETAILED DESCRIPTION:
Patients meeting inclusion criteria would be randomised after admission. Those patients in experimental arm shall receive the TAP block under USG guidance while those in control arm do not receive any block. Surgery shall be proceeded in the usual manner in all the patients and assessment for pain starts in the immediate post operative or recovery room after the patient is completely conscious. The total amount of analgesic required by the patient is measured. Pain assessment is done using the visual analog scale (VAS) at regular intervals until follow up review.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing laparoscopic ventral hernia repair during the study period

Exclusion Criteria:

* Age <15 or greater than 75 years
* ASA > 3
* Obstructed , recurrent or strangulated hernia
* Lap assisted open hernia repair
* Patients undergoing component separation
* Parastomal hernia, spigelian hernia, lumbar hernia
* Patients with Chronic kidney disease, bronchial asthma
* Patients allergic to bupivacaine or NSAIDs
* Not willing to participate

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Post operative cumulative analgesic requirement | 24 hours after surgery
  The amount of analgesic required by the patient during hospital stay

SECONDARY OUTCOMES:
Post-operative hospital stay | 7 days from primary surgery
  The time taken to get discharged from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: C C Palanivelu, MS, MCh, Principal Investigator — Gem Hospital and research center
Locations (1):
- Gem hospital and research centre, Coimbatore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No